CLINICAL TRIAL: NCT05282277
Title: Examining the Effects of Estradiol on Neural and Molecular Response to Rewards in Perimenopausal-Onset Anhedonia and Psychosis
Brief Title: Examining the Effects of Estradiol on Neural and Molecular Response to Reward
Acronym: PEEPS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-2230; R01MH128238-01 (NIH)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Depression; Psychosis; Anhedonia
Keywords: Reproductive Affective Disorder; Anhedonia; Perimenopause; Estrogen; Hormone Replacement Therapy; Mood Disorders; Estradiol Treatment; Sex Steroids; Psychosis Symptoms; Depressive Disorders; Estradiol; Hormones; Reward Activation; Reproductive Control Agents
MeSH Terms: conditions — Depression; Psychotic Disorders; Anhedonia; Mood Disorders; Depressive Disorder | interventions — Estradiol; Progesterone; Raclopride

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized placebo-controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Perimenopausal women with mild-to-moderate anhedonia + absent-to-mild psychosis, active group (Experimental): Participants will be randomly assigned to take 100 μg/day of transdermal estradiol for 3 weeks followed by 1 week of combined 100 μg/day of transdermal estradiol and 200 mg/day progesterone.
  Interventions: Drug: Transdermal Estradiol; Drug: Micronized Progesterone; Drug: Raclopride C11
- Perimenopausal women with mild-to-moderate anhedonia + absent-to-mild psychosis, placebo group (Experimental): Participants will be randomly assigned to receive a matching placebo patch for 3 weeks.
  Interventions: Drug: Matching Placebo Patch; Drug: Raclopride C11
- Perimenopausal women with mild-to-moderate anhedonia + moderate psychosis, active group (Experimental): Participants will be randomly assigned to take 100 μg/day of transdermal estradiol for 3 weeks followed by 1 week of combined 100 μg/day of transdermal estradiol and 200 mg/day progesterone.
  Interventions: Drug: Transdermal Estradiol; Drug: Micronized Progesterone; Drug: Raclopride C11
- Perimenopausal women with mild-to-moderate anhedonia + moderate psychosis, placebo group (Experimental): Participants will be randomly assigned to receive a matching placebo patch for 3 weeks.
  Interventions: Drug: Matching Placebo Patch; Drug: Raclopride C11
- Perimenopausal women with high anhedonia + absent-to-mild psychosis, active group (Experimental): Participants will be randomly assigned to take 100 μg/day of transdermal estradiol for 3 weeks followed by 1 week of combined 100 μg/day of transdermal estradiol and 200 mg/day progesterone.
  Interventions: Drug: Transdermal Estradiol; Drug: Micronized Progesterone; Drug: Raclopride C11
- Perimenopausal women with high anhedonia + absent-to-mild psychosis, placebo group (Experimental): Participants will be randomly assigned to receive a matching placebo patch for 3 weeks.
  Interventions: Drug: Matching Placebo Patch; Drug: Raclopride C11
- Perimenopausal women with high anhedonia + moderate psychosis, active group (Experimental): Participants will be randomly assigned to take 100 μg/day of transdermal estradiol for 3 weeks followed by 1 week of combined 100 μg/day of transdermal estradiol and 200 mg/day progesterone.
  Interventions: Drug: Transdermal Estradiol; Drug: Micronized Progesterone; Drug: Raclopride C11
- Perimenopausal women with high anhedonia + moderate psychosis, placebo group (Experimental): Participants will be randomly assigned to receive a matching placebo patch for 3 weeks.
  Interventions: Drug: Matching Placebo Patch; Drug: Raclopride C11

INTERVENTIONS:
Drug: Transdermal Estradiol — Participants will be randomized to receive transdermal estradiol (100μg/day) patch for 3 weeks.
  Other Names: Climara
  Arms: Perimenopausal women with high anhedonia + absent-to-mild psychosis, active group; Perimenopausal women with high anhedonia + moderate psychosis, active group; Perimenopausal women with mild-to-moderate anhedonia + absent-to-mild psychosis, active group; Perimenopausal women with mild-to-moderate anhedonia + moderate psychosis, active group
Drug: Micronized Progesterone — Participants will receive an additional week of micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
  Other Names: Prometrium
  Arms: Perimenopausal women with high anhedonia + absent-to-mild psychosis, active group; Perimenopausal women with high anhedonia + moderate psychosis, active group; Perimenopausal women with mild-to-moderate anhedonia + absent-to-mild psychosis, active group; Perimenopausal women with mild-to-moderate anhedonia + moderate psychosis, active group
Drug: Matching Placebo Patch — Participants will be randomized to receive a transdermal estradiol-matching placebo patch for 3 weeks
  Other Names: Placebo
  Arms: Perimenopausal women with high anhedonia + absent-to-mild psychosis, placebo group; Perimenopausal women with high anhedonia + moderate psychosis, placebo group; Perimenopausal women with mild-to-moderate anhedonia + absent-to-mild psychosis, placebo group; Perimenopausal women with mild-to-moderate anhedonia + moderate psychosis, placebo group
Drug: Raclopride C11 — All Participants will receive two PET-MR scans using [11C]raclopride IV as the tracer. The first scan will occur at baseline and the second at post treatment after 3 weeks.
  Other Names: [C11]Raclopride

SUMMARY:
This proposal will examine the effects of estradiol administration on perimenopausal-onset (PO) anhedonia and psychosis symptoms as well as on brain function using simultaneous positron emission tomography and functional magnetic resonance imaging (PET-MR).

DETAILED DESCRIPTION:
The transition to menopause (the "perimenopause") is characterized by increased risk for new onset of depression and psychosis. Our work and that of others has demonstrated that a prominent symptom of perimenopausal-onset (PO) depression is anhedonia, contributing significantly to distress and functional impairment. Additionally, the incidence of psychosis in women may increase during this period. Declining or low levels of estradiol, particularly in the late perimenopause, may play a role in the pathogenesis of PO anhedonia and PO psychosis via effects on mesolimbic brain reward circuitry and dopamine (DA) neurotransmission. Preclinical evidence has established that estradiol modulates dopamine systems and reward-related behaviors and estradiol withdrawal evokes loss of dopaminergic functions. Whereas estrogen therapy has shown benefits in reducing mood and psychotic symptoms in perimenopausal women, no study has examined the neural mechanisms underlying such effects in a transdiagnostic sample.

This project will examine the effects of estradiol administration on perimenopausal-onset (PO) anhedonia and psychosis using simultaneous positron emission tomography and functional magnetic resonance imaging (PET-MR). Preliminary data presented here demonstrate that anhedonia is associated with decreased striatal DA release to rewards using PET with the D2/D3 DA receptor antagonist [11C]raclopride; anhedonia and psychosis are characterized by altered striatal activation to rewards using fMRI; estradiol impacts neural responses to rewards in PO anhedonia and PO psychosis; and estradiol improves PO anhedonia and PO psychosis. This project proposes to extend these lines of research by using simultaneous PET-MR to investigate the effects of transdermal estradiol, administered as a mechanistic probe, on PO anhedonia and PO psychosis in a transdiagnostic sample of women using a double-blind between-groups placebo-controlled design. This sample will be enriched for anhedonia (i.e., at least mild anhedonia). Although anhedonia and psychosis will be analyzed dimensionally, our recruitment and stratification strategy will ensure that a range of symptom severities (mild-to-moderate or high PO anhedonia; absent-to-mild or moderate PO psychosis) are equally balanced and randomized to each experimental group (estradiol or placebo). Our central hypotheses are that the mesolimbic DA system is impaired in PO anhedonia and psychosis, that estradiol administration will normalize neural responses to rewards (measured by fMRI) and striatal DA functioning (measured by PET), and that the degree of change in striatal functioning will be associated with the degree of change in PO anhedonia and PO psychosis.

Specific Aim 1 (baseline associations between PO anhedonia, PO psychosis, and PET-MR): Characterize, at baseline, associations between PO anhedonia and PO psychosis symptom severity and reward-related striatal activation measured by fMRI, and tonic and phasic striatal DA activity measured by [11C]raclopride PET.

Specific Aim 2 (estradiol effects on PO anhedonia and PET-MR): Determine the effects of estradiol (vs. placebo) on PO anhedonia and changes in PET-MR metrics related to reward processing.

Specific Aim 3 (estradiol effects on PO psychosis and PET-MR): Determine the effects of estradiol (vs. placebo) on PO psychosis and changes in PET-MR metrics related to reward processing.

This project will improve our understanding of PO anhedonia and psychosis and the mechanisms of action of the effect of estradiol on PO anhedonia and psychosis. This research will provide new mechanistic endpoints to evaluate novel PO anhedonia and psychosis treatments that target the mesolimbic DA system.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures, lifestyle considerations, and availability for the duration of the study
* 44-55 years old unmedicated perimenopausal women who have ≥ 2 skipped menstrual cycles, amenorrhea ≥ 60 days, corresponding to the late menopause transition (Stages of Reproductive Aging Workshop (STRAW stage -1).
* Anhedonia or psychosis symptoms that began during the period of menstrual irregularity.
* Clinician's Global Impression Scale-Severity score (CGI-S) > 3 to confirm a clinically impaired sample.
* Anhedonia severity inclusion criteria and stratification: All participants will have Snaith-Hamilton Pleasure Scale (SHAPS) scores > 20 consistent with the NIMH Fast-Fail Trial for Mood and Anxiety Disorders, corresponding to clinically impairing anhedonia.
* Psychosis severity inclusion criteria and stratification: Participants will be stratified according to scores on the psychotic subscale of the Brief Psychiatric Rating Scale (BPRS)
* Willingness to adhere to the estradiol regimen

Exclusion Criteria:

* Pregnancy; allergies to any active or inactive ingredients in the Climara® patch or Prometrium®.
* BMI < 18 or > 35 kg/m^2
* A history of chronic menstrual cycle irregularity, meaning > 1 year without menses
* MR contraindications: Metal in the body, dental work other than fillings or gold, tattoos, metal injury, any other implant unless they are 100% plastic.
* PET contradictions: participation in >1 research study in the past 12 months that included ionizing radiation exceeding 3 rem to the whole body (e.g., PET, CT). Standard of care imaging is not exclusionary.
* The use of psychotropics or hormonal preparations.
* History of psychiatric illness during the 2 years before the onset of perimenopause.
* History of chronic, recurrent mood or psychotic disorders (i.e., more than one non-reproductive-related mood episode prior to the perimenopausal index episode).
* A history of mood episodes requiring hospitalization.
* Current mania;
* Depressive episode(s) within 2 years of enrollment not associated with the transition to menopause;
* A history of suicide attempts within the last year or current active suicidal ideation with intent and plan.
* Neurological conditions (e.g., history of seizure or TBI)
* Brain stimulation treatment in the past six months.
* Endometriosis;
* First degree relative with premenopausal breast cancer or breast cancer presenting in both breasts or multiple family members (greater than three relatives) with postmenopausal breast cancer.
* Current medication use (i.e., current psychotropics, current anti-hypertensives, current statins, current hormonal preparations, or frequent use of anti-inflammatory agents (> 10 times/month)). Women will be allowed to enroll who take medications without known mood effects (e.g. stable thyroid hormone replacement and occasional (< 5 times/month) use of Ambien)*;
* Pregnant, breastfeeding or trying to conceive;
* Last menstrual period more than 12 months prior to enrollment;
* History of undiagnosed vaginal bleeding;
* Undiagnosed enlargement of the ovaries;
* Polycystic ovary syndrome;
* History of breast or ovarian cancer;
* First degree relative with ovarian cancer;
* Abnormal finding in a provider breast exam and/or mammogram;
* Known carrier of BRCA1 or 2 mutation;
* Porphyria;
* Malignant melanoma;
* Hodgkin's disease;
* Recurrent migraine headaches that are preceded by aura;
* Gallbladder or pancreatic disease**;
* Heart or kidney disease**;
* Liver disease;
* cerebrovascular disease (stroke);
* First degree relative with history of heart attack or stroke;
* Current nicotine use;
* Self-reported claustrophobia
* Peanut allergy

  * all reported prescription medications will be reviewed and cleared by a study physician prior to a participant's enrollment;

    * participants will be given the opportunity to describe these conditions in the online screening survey. Reported conditions that are acute in nature and/or benign will be reviewed by a study physician and exclusions will be decided case-by-case. All chronic conditions will be exclusionary. For those where it is deemed that an exclusion does not apply, primary analyses will not be affected, but exploratory analyses will be conducted excluding these individuals

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Striatal Activation Between Groups during the MID task | Baseline (week 3) to Endpoint (week 7)
  Characterize reward-related striatal activation measured by fMRI using the Monetary Incentive Delay (MID) task to elicit blood-oxygen-level dependent (BOLD) responses. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) response to win trials versus non-win trials. Reactivity is then compared between the two groups.

SECONDARY OUTCOMES:
Changes in PO Psychosis Symptoms following Estradiol Administration Using the BPRS | Baseline (week 3) to Endpoint (week 7)
  Determine the effects of estradiol (vs. placebo) on PO psychosis symptoms using the Brief Psychiatric Rating Scale (BPRS).The BPRS is an 18-item clinician rated psychosis measure that examines the severity of psychotic symptoms. Individuals with psychotic major depression typically have BPRS positive symptom subscale scores 7-11, and a score of 6 best differentiates psychotic MDD from nonpsychotic MDD.
Changes in PO Anhedonia Following Estradiol Administration Using the SHAPS | Baseline (week 3) to Endpoint (week 7)
  Determine the effects of estradiol (vs. placebo) on PO anhedonia symptoms using the Snaith-Hamilton Pleasure Scale (SHAPS). The SHAPS is a 14-item self-rated anhedonia scale. Items are comprised of statements that participants rate as "strongly disagree" (1), "disagree" (2), "agree" (3), or "strongly agree" (4). The lowest possible score is 14, the highest possible score is 56 (greatest anhedonia)
Change in striatal phasic DA release and background DA tone to rewards measured by [11C]raclopride PET using the Monetary Incentive Delay (MID) task. | Baseline (week 3) to Endpoint (week 7)
  Binding potential changes due to DA release and competition will be determined using a dynamic occupancy model. We will use baseline nondisplaceable binding potential (BPND) and change in BPND following task onset (ΔBPND%) to determine differences between groups in terms of the baseline (tonic) state and the activation (phasic) state.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal E Schiller, PhD, Principal Investigator — UNC School of Medicine - Department of Psychiatry; Gabriel Dichter, PhD, Principal Investigator — UNC School of Medicine - CIDD
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication.
Access Criteria: Approval from an IRB, IEC, or REB, as applicable and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Bromberger JT, Matthews KA, Schott LL, Brockwell S, Avis NE, Kravitz HM, Everson-Rose SA, Gold EB, Sowers M, Randolph JF Jr. Depressive symptoms during the menopausal transition: the Study of Women's Health Across the Nation (SWAN). J Affect Disord. 2007 Nov;103(1-3):267-72. doi: 10.1016/j.jad.2007.01.034. Epub 2007 Feb 28. PMID 17331589
- [Background] Freeman EW, Sammel MD, Boorman DW, Zhang R. Longitudinal pattern of depressive symptoms around natural menopause. JAMA Psychiatry. 2014 Jan;71(1):36-43. doi: 10.1001/jamapsychiatry.2013.2819. PMID 24227182
- [Background] Maki PM, Kornstein SG, Joffe H, Bromberger JT, Freeman EW, Athappilly G, Bobo WV, Rubin LH, Koleva HK, Cohen LS, Soares CN. Guidelines for the Evaluation and Treatment of Perimenopausal Depression: Summary and Recommendations. J Womens Health (Larchmt). 2019 Feb;28(2):117-134. doi: 10.1089/jwh.2018.27099.mensocrec. Epub 2018 Sep 5. PMID 30182804
- [Background] Frokjaer VG. Pharmacological sex hormone manipulation as a risk model for depression. J Neurosci Res. 2020 Jul;98(7):1283-1292. doi: 10.1002/jnr.24632. Epub 2020 May 12. PMID 32399989
- [Background] Schiller CE, Johnson SL, Abate AC, Schmidt PJ, Rubinow DR. Reproductive Steroid Regulation of Mood and Behavior. Compr Physiol. 2016 Jun 13;6(3):1135-60. doi: 10.1002/cphy.c150014. PMID 27347888
- [Background] Dichter GS, Damiano CA, Allen JA. Reward circuitry dysfunction in psychiatric and neurodevelopmental disorders and genetic syndromes: animal models and clinical findings. J Neurodev Disord. 2012 Jul 6;4(1):19. doi: 10.1186/1866-1955-4-19. PMID 22958744
- [Background] Nusslock R, Alloy LB. Reward processing and mood-related symptoms: An RDoC and translational neuroscience perspective. J Affect Disord. 2017 Jul;216:3-16. doi: 10.1016/j.jad.2017.02.001. Epub 2017 Feb 4. PMID 28237133
- [Background] Macoveanu J, Meluken I, Chase HW, Phillips ML, Kessing LV, Siebner HR, Vinberg M, Miskowiak KW. Reduced frontostriatal response to expected value and reward prediction error in remitted monozygotic twins with mood disorders and their unaffected high-risk co-twins. Psychol Med. 2021 Jul;51(10):1637-1646. doi: 10.1017/S0033291720000367. Epub 2020 Mar 2. PMID 32115012
- [Background] Guffanti G, Kumar P, Admon R, Treadway MT, Hall MH, Mehta M, Douglas S, Arulpragasam AR, Pizzagalli DA. Depression genetic risk score is associated with anhedonia-related markers across units of analysis. Transl Psychiatry. 2019 Sep 19;9(1):236. doi: 10.1038/s41398-019-0566-7. PMID 31537779
- [Background] Kumar P, Goer F, Murray L, Dillon DG, Beltzer ML, Cohen AL, Brooks NH, Pizzagalli DA. Impaired reward prediction error encoding and striatal-midbrain connectivity in depression. Neuropsychopharmacology. 2018 Jun;43(7):1581-1588. doi: 10.1038/s41386-018-0032-x. Epub 2018 Feb 26. PMID 29540863
- [Background] Treadway MT, Zald DH. Reconsidering anhedonia in depression: lessons from translational neuroscience. Neurosci Biobehav Rev. 2011 Jan;35(3):537-55. doi: 10.1016/j.neubiorev.2010.06.006. Epub 2010 Jul 11. PMID 20603146
- [Background] Willner P, Scheel-Kruger J, Belzung C. The neurobiology of depression and antidepressant action. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 1):2331-71. doi: 10.1016/j.neubiorev.2012.12.007. Epub 2012 Dec 19. PMID 23261405
- [Background] Pizzagalli DA. Depression, stress, and anhedonia: toward a synthesis and integrated model. Annu Rev Clin Psychol. 2014;10:393-423. doi: 10.1146/annurev-clinpsy-050212-185606. PMID 24471371
- [Background] Hamilton JP, Sacchet MD, Hjornevik T, Chin FT, Shen B, Kampe R, Park JH, Knutson BD, Williams LM, Borg N, Zaharchuk G, Camacho MC, Mackey S, Heilig M, Drevets WC, Glover GH, Gambhir SS, Gotlib IH. Striatal dopamine deficits predict reductions in striatal functional connectivity in major depression: a concurrent 11C-raclopride positron emission tomography and functional magnetic resonance imaging investigation. Transl Psychiatry. 2018 Nov 30;8(1):264. doi: 10.1038/s41398-018-0316-2. PMID 30504860
- [Background] Treadway MT. The Neurobiology of Motivational Deficits in Depression--An Update on Candidate Pathomechanisms. Curr Top Behav Neurosci. 2016;27:337-55. doi: 10.1007/7854_2015_400. PMID 26475160
- [Background] Whitton AE, Treadway MT, Pizzagalli DA. Reward processing dysfunction in major depression, bipolar disorder and schizophrenia. Curr Opin Psychiatry. 2015 Jan;28(1):7-12. doi: 10.1097/YCO.0000000000000122. PMID 25415499
- [Background] Howes OD, Kapur S. The dopamine hypothesis of schizophrenia: version III--the final common pathway. Schizophr Bull. 2009 May;35(3):549-62. doi: 10.1093/schbul/sbp006. Epub 2009 Mar 26. PMID 19325164
- [Background] Morris RW, Vercammen A, Lenroot R, Moore L, Langton JM, Short B, Kulkarni J, Curtis J, O'Donnell M, Weickert CS, Weickert TW. Disambiguating ventral striatum fMRI-related BOLD signal during reward prediction in schizophrenia. Mol Psychiatry. 2012 Mar;17(3):235, 280-9. doi: 10.1038/mp.2011.75. Epub 2011 Jun 28. PMID 21709684
- [Background] Morris R, Griffiths O, Le Pelley ME, Weickert TW. Attention to irrelevant cues is related to positive symptoms in schizophrenia. Schizophr Bull. 2013 May;39(3):575-82. doi: 10.1093/schbul/sbr192. Epub 2012 Jan 20. PMID 22267535
- [Background] Wotruba D, Heekeren K, Michels L, Buechler R, Simon JJ, Theodoridou A, Kollias S, Rossler W, Kaiser S. Symptom dimensions are associated with reward processing in unmedicated persons at risk for psychosis. Front Behav Neurosci. 2014 Nov 18;8:382. doi: 10.3389/fnbeh.2014.00382. eCollection 2014. PMID 25477792
- [Background] van Timmeren T, Quail SL, Balleine BW, Geurts DEM, Goudriaan AE, van Holst RJ. Intact corticostriatal control of goal-directed action in Alcohol Use Disorder: a Pavlovian-to-instrumental transfer and outcome-devaluation study. Sci Rep. 2020 Mar 18;10(1):4949. doi: 10.1038/s41598-020-61892-5. PMID 32188908
- [Background] Kirschner M, Hager OM, Muff L, Bischof M, Hartmann-Riemer MN, Kluge A, Habermeyer B, Seifritz E, Tobler PN, Kaiser S. Ventral Striatal Dysfunction and Symptom Expression in Individuals With Schizotypal Personality Traits and Early Psychosis. Schizophr Bull. 2018 Jan 13;44(1):147-157. doi: 10.1093/schbul/sbw142. PMID 27798223
- [Background] Romaniuk L, Honey GD, King JR, Whalley HC, McIntosh AM, Levita L, Hughes M, Johnstone EC, Day M, Lawrie SM, Hall J. Midbrain activation during Pavlovian conditioning and delusional symptoms in schizophrenia. Arch Gen Psychiatry. 2010 Dec;67(12):1246-54. doi: 10.1001/archgenpsychiatry.2010.169. PMID 21135324
- [Background] Roiser JP, Howes OD, Chaddock CA, Joyce EM, McGuire P. Neural and behavioral correlates of aberrant salience in individuals at risk for psychosis. Schizophr Bull. 2013 Nov;39(6):1328-36. doi: 10.1093/schbul/sbs147. Epub 2012 Dec 12. PMID 23236077
- [Background] Modinos G, Tseng HH, Falkenberg I, Samson C, McGuire P, Allen P. Neural correlates of aberrant emotional salience predict psychotic symptoms and global functioning in high-risk and first-episode psychosis. Soc Cogn Affect Neurosci. 2015 Oct;10(10):1429-36. doi: 10.1093/scan/nsv035. Epub 2015 Mar 25. PMID 25809400
- [Background] Jensen J, Willeit M, Zipursky RB, Savina I, Smith AJ, Menon M, Crawley AP, Kapur S. The formation of abnormal associations in schizophrenia: neural and behavioral evidence. Neuropsychopharmacology. 2008 Feb;33(3):473-9. doi: 10.1038/sj.npp.1301437. Epub 2007 May 2. PMID 17473838
- [Background] Laruelle M, Abi-Dargham A. Dopamine as the wind of the psychotic fire: new evidence from brain imaging studies. J Psychopharmacol. 1999 Dec;13(4):358-71. doi: 10.1177/026988119901300405. PMID 10667612
- [Background] van Winkel R, Stefanis NC, Myin-Germeys I. Psychosocial stress and psychosis. A review of the neurobiological mechanisms and the evidence for gene-stress interaction. Schizophr Bull. 2008 Nov;34(6):1095-105. doi: 10.1093/schbul/sbn101. Epub 2008 Aug 20. PMID 18718885
- [Background] Cannon TD, van Erp TG, Bearden CE, Loewy R, Thompson P, Toga AW, Huttunen MO, Keshavan MS, Seidman LJ, Tsuang MT. Early and late neurodevelopmental influences in the prodrome to schizophrenia: contributions of genes, environment, and their interactions. Schizophr Bull. 2003;29(4):653-69. doi: 10.1093/oxfordjournals.schbul.a007037. PMID 14989405
- [Background] Howes OD, McDonald C, Cannon M, Arseneault L, Boydell J, Murray RM. Pathways to schizophrenia: the impact of environmental factors. Int J Neuropsychopharmacol. 2004 Mar;7 Suppl 1:S7-S13. doi: 10.1017/S1461145704004122. PMID 14972079
- [Background] Maia TV, Frank MJ. An Integrative Perspective on the Role of Dopamine in Schizophrenia. Biol Psychiatry. 2017 Jan 1;81(1):52-66. doi: 10.1016/j.biopsych.2016.05.021. Epub 2016 Jun 1. PMID 27452791
- [Background] Frank MJ. Dynamic dopamine modulation in the basal ganglia: a neurocomputational account of cognitive deficits in medicated and nonmedicated Parkinsonism. J Cogn Neurosci. 2005 Jan;17(1):51-72. doi: 10.1162/0898929052880093. PMID 15701239
- [Background] Gerfen CR, Surmeier DJ. Modulation of striatal projection systems by dopamine. Annu Rev Neurosci. 2011;34:441-66. doi: 10.1146/annurev-neuro-061010-113641. PMID 21469956
- [Background] Brown JK, Waltz JA, Strauss GP, McMahon RP, Frank MJ, Gold JM. Hypothetical decision making in schizophrenia: the role of expected value computation and "irrational" biases. Psychiatry Res. 2013 Sep 30;209(2):142-9. doi: 10.1016/j.psychres.2013.02.034. Epub 2013 May 9. PMID 23664664
- [Background] Strauss GP, Robinson BM, Waltz JA, Frank MJ, Kasanova Z, Herbener ES, Gold JM. Patients with schizophrenia demonstrate inconsistent preference judgments for affective and nonaffective stimuli. Schizophr Bull. 2011 Nov;37(6):1295-304. doi: 10.1093/schbul/sbq047. Epub 2010 May 19. PMID 20484522
- [Background] Howes OD, Kambeitz J, Kim E, Stahl D, Slifstein M, Abi-Dargham A, Kapur S. The nature of dopamine dysfunction in schizophrenia and what this means for treatment. Arch Gen Psychiatry. 2012 Aug;69(8):776-86. doi: 10.1001/archgenpsychiatry.2012.169. PMID 22474070
- [Background] Abi-Dargham A, Gil R, Krystal J, Baldwin RM, Seibyl JP, Bowers M, van Dyck CH, Charney DS, Innis RB, Laruelle M. Increased striatal dopamine transmission in schizophrenia: confirmation in a second cohort. Am J Psychiatry. 1998 Jun;155(6):761-7. doi: 10.1176/ajp.155.6.761. PMID 9619147
- [Background] Breier A, Su TP, Saunders R, Carson RE, Kolachana BS, de Bartolomeis A, Weinberger DR, Weisenfeld N, Malhotra AK, Eckelman WC, Pickar D. Schizophrenia is associated with elevated amphetamine-induced synaptic dopamine concentrations: evidence from a novel positron emission tomography method. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2569-74. doi: 10.1073/pnas.94.6.2569. PMID 9122236
- [Background] Kestler LP, Walker E, Vega EM. Dopamine receptors in the brains of schizophrenia patients: a meta-analysis of the findings. Behav Pharmacol. 2001 Sep;12(5):355-71. doi: 10.1097/00008877-200109000-00007. PMID 11710751
- [Background] Laruelle M, Abi-Dargham A, van Dyck CH, Gil R, D'Souza CD, Erdos J, McCance E, Rosenblatt W, Fingado C, Zoghbi SS, Baldwin RM, Seibyl JP, Krystal JH, Charney DS, Innis RB. Single photon emission computerized tomography imaging of amphetamine-induced dopamine release in drug-free schizophrenic subjects. Proc Natl Acad Sci U S A. 1996 Aug 20;93(17):9235-40. doi: 10.1073/pnas.93.17.9235. PMID 8799184
- [Background] Hietala J, Syvalahti E, Vuorio K, Rakkolainen V, Bergman J, Haaparanta M, Solin O, Kuoppamaki M, Kirvela O, Ruotsalainen U, et al. Presynaptic dopamine function in striatum of neuroleptic-naive schizophrenic patients. Lancet. 1995 Oct 28;346(8983):1130-1. doi: 10.1016/s0140-6736(95)91801-9. PMID 7475604
- [Background] Hietala J, Syvalahti E, Vilkman H, Vuorio K, Rakkolainen V, Bergman J, Haaparanta M, Solin O, Kuoppamaki M, Eronen E, Ruotsalainen U, Salokangas RK. Depressive symptoms and presynaptic dopamine function in neuroleptic-naive schizophrenia. Schizophr Res. 1999 Jan 4;35(1):41-50. doi: 10.1016/s0920-9964(98)00113-3. PMID 9988840
- [Background] Howes OD, Montgomery AJ, Asselin MC, Murray RM, Valli I, Tabraham P, Bramon-Bosch E, Valmaggia L, Johns L, Broome M, McGuire PK, Grasby PM. Elevated striatal dopamine function linked to prodromal signs of schizophrenia. Arch Gen Psychiatry. 2009 Jan;66(1):13-20. doi: 10.1001/archgenpsychiatry.2008.514. PMID 19124684
- [Background] Lindstrom LH, Gefvert O, Hagberg G, Lundberg T, Bergstrom M, Hartvig P, Langstrom B. Increased dopamine synthesis rate in medial prefrontal cortex and striatum in schizophrenia indicated by L-(beta-11C) DOPA and PET. Biol Psychiatry. 1999 Sep 1;46(5):681-8. doi: 10.1016/s0006-3223(99)00109-2. PMID 10472420
- [Background] Howes OD, Montgomery AJ, Asselin MC, Murray RM, Grasby PM, McGuire PK. Molecular imaging studies of the striatal dopaminergic system in psychosis and predictions for the prodromal phase of psychosis. Br J Psychiatry Suppl. 2007 Dec;51:s13-8. doi: 10.1192/bjp.191.51.s13. PMID 18055930
- [Background] Steinberg EM, Rubinow DR, Bartko JJ, Fortinsky PM, Haq N, Thompson K, Schmidt PJ. A cross-sectional evaluation of perimenopausal depression. J Clin Psychiatry. 2008 Jun;69(6):973-80. doi: 10.4088/jcp.v69n0614. PMID 18505304
- [Background] Schmidt PJ, Nieman L, Danaceau MA, Tobin MB, Roca CA, Murphy JH, Rubinow DR. Estrogen replacement in perimenopause-related depression: a preliminary report. Am J Obstet Gynecol. 2000 Aug;183(2):414-20. doi: 10.1067/mob.2000.106004. PMID 10942479
- [Background] The NAMS 2017 Hormone Therapy Position Statement Advisory Panel. The 2017 hormone therapy position statement of The North American Menopause Society. Menopause. 2017 Jul;24(7):728-753. doi: 10.1097/GME.0000000000000921. PMID 28650869
- [Background] Kulkarni J, Gavrilidis E, Wang W, Worsley R, Fitzgerald PB, Gurvich C, Van Rheenen T, Berk M, Burger H. Estradiol for treatment-resistant schizophrenia: a large-scale randomized-controlled trial in women of child-bearing age. Mol Psychiatry. 2015 Jun;20(6):695-702. doi: 10.1038/mp.2014.33. Epub 2014 Apr 15. PMID 24732671
- [Background] Burger H. The menopausal transition--endocrinology. J Sex Med. 2008 Oct;5(10):2266-73. doi: 10.1111/j.1743-6109.2008.00921.x. Epub 2008 Jul 1. PMID 18624962
- [Background] Fink G, Sumner BE, Rosie R, Grace O, Quinn JP. Estrogen control of central neurotransmission: effect on mood, mental state, and memory. Cell Mol Neurobiol. 1996 Jun;16(3):325-44. doi: 10.1007/BF02088099. PMID 8818400
- [Background] Barth C, Villringer A, Sacher J. Sex hormones affect neurotransmitters and shape the adult female brain during hormonal transition periods. Front Neurosci. 2015 Feb 20;9:37. doi: 10.3389/fnins.2015.00037. eCollection 2015. PMID 25750611
- [Background] Gupta R, Assalman I, Bottlender R. Menopause and schizophrenia. Menopause Int. 2012 Mar;18(1):10-4. doi: 10.1258/mi.2012.011116. Epub 2012 Feb 3. PMID 22308532
- [Background] Euvrard C, Oberlander C, Boissier JR. Antidopaminergic effect of estrogens at the striatal level. J Pharmacol Exp Ther. 1980 Jul;214(1):179-85. PMID 7391967
- [Background] Di Paolo T, Rouillard C, Bedard P. 17 beta-Estradiol at a physiological dose acutely increases dopamine turnover in rat brain. Eur J Pharmacol. 1985 Nov 5;117(2):197-203. doi: 10.1016/0014-2999(85)90604-1. PMID 4076343
- [Background] Thompson TL, Moss RL. Estrogen regulation of dopamine release in the nucleus accumbens: genomic- and nongenomic-mediated effects. J Neurochem. 1994 May;62(5):1750-6. doi: 10.1046/j.1471-4159.1994.62051750.x. PMID 8158125
- [Background] Calipari ES, Juarez B, Morel C, Walker DM, Cahill ME, Ribeiro E, Roman-Ortiz C, Ramakrishnan C, Deisseroth K, Han MH, Nestler EJ. Dopaminergic dynamics underlying sex-specific cocaine reward. Nat Commun. 2017 Jan 10;8:13877. doi: 10.1038/ncomms13877. PMID 28072417
- [Background] Shams WM, Cossette MP, Shizgal P, Brake WG. 17beta-estradiol locally increases phasic dopamine release in the dorsal striatum. Neurosci Lett. 2018 Feb 5;665:29-32. doi: 10.1016/j.neulet.2017.11.039. Epub 2017 Nov 22. PMID 29175028
- [Background] Madularu D, Kulkarni P, Yee JR, Kenkel WM, Shams WM, Ferris CF, Brake WG. High estrogen and chronic haloperidol lead to greater amphetamine-induced BOLD activation in awake, amphetamine-sensitized female rats. Horm Behav. 2016 Jun;82:56-63. doi: 10.1016/j.yhbeh.2016.04.007. Epub 2016 May 15. PMID 27154458
- [Background] Frank TC, Kim GL, Krzemien A, Van Vugt DA. Effect of menstrual cycle phase on corticolimbic brain activation by visual food cues. Brain Res. 2010 Dec 2;1363:81-92. doi: 10.1016/j.brainres.2010.09.071. Epub 2010 Oct 25. PMID 20920491
- [Background] Ossewaarde L, van Wingen GA, Rijpkema M, Backstrom T, Hermans EJ, Fernandez G. Menstrual cycle-related changes in amygdala morphology are associated with changes in stress sensitivity. Hum Brain Mapp. 2013 May;34(5):1187-93. doi: 10.1002/hbm.21502. Epub 2011 Dec 8. PMID 22162177
- [Background] Bayer J, Bandurski P, Sommer T. Differential modulation of activity related to the anticipation of monetary gains and losses across the menstrual cycle. Eur J Neurosci. 2013 Nov;38(10):3519-26. doi: 10.1111/ejn.12347. Epub 2013 Aug 25. PMID 23981052
- [Background] Dreher JC, Schmidt PJ, Kohn P, Furman D, Rubinow D, Berman KF. Menstrual cycle phase modulates reward-related neural function in women. Proc Natl Acad Sci U S A. 2007 Feb 13;104(7):2465-70. doi: 10.1073/pnas.0605569104. Epub 2007 Jan 31. PMID 17267613
- [Background] Reimers L, Buchel C, Diekhof EK. How to be patient. The ability to wait for a reward depends on menstrual cycle phase and feedback-related activity. Front Neurosci. 2014 Dec 9;8:401. doi: 10.3389/fnins.2014.00401. eCollection 2014. PMID 25538555
- [Background] Diekhof EK, Ratnayake M. Menstrual cycle phase modulates reward sensitivity and performance monitoring in young women: Preliminary fMRI evidence. Neuropsychologia. 2016 Apr;84:70-80. doi: 10.1016/j.neuropsychologia.2015.10.016. Epub 2015 Oct 22. PMID 26471712
- [Background] Thomas J, Metereau E, Dechaud H, Pugeat M, Dreher JC. Hormonal treatment increases the response of the reward system at the menopause transition: a counterbalanced randomized placebo-controlled fMRI study. Psychoneuroendocrinology. 2014 Dec;50:167-80. doi: 10.1016/j.psyneuen.2014.08.012. Epub 2014 Sep 1. PMID 25222702
- [Background] Becker JB. Estrogen rapidly potentiates amphetamine-induced striatal dopamine release and rotational behavior during microdialysis. Neurosci Lett. 1990 Oct 16;118(2):169-71. doi: 10.1016/0304-3940(90)90618-j. PMID 2125712
- [Background] Inagaki T, Gautreaux C, Luine V. Acute estrogen treatment facilitates recognition memory consolidation and alters monoamine levels in memory-related brain areas. Horm Behav. 2010 Aug;58(3):415-26. doi: 10.1016/j.yhbeh.2010.05.013. Epub 2010 May 27. PMID 20553724
- [Background] Bayer J, Rusch T, Zhang L, Glascher J, Sommer T. Dose-dependent effects of estrogen on prediction error related neural activity in the nucleus accumbens of healthy young women. Psychopharmacology (Berl). 2020 Mar;237(3):745-755. doi: 10.1007/s00213-019-05409-7. Epub 2019 Nov 26. PMID 31773208
- [Background] Gogos A, Sbisa AM, Sun J, Gibbons A, Udawela M, Dean B. A Role for Estrogen in Schizophrenia: Clinical and Preclinical Findings. Int J Endocrinol. 2015;2015:615356. doi: 10.1155/2015/615356. Epub 2015 Sep 27. PMID 26491441
- [Background] Seeman P. Targeting the dopamine D2 receptor in schizophrenia. Expert Opin Ther Targets. 2006 Aug;10(4):515-31. doi: 10.1517/14728222.10.4.515. PMID 16848689
- [Background] Seeman P. Dopamine D2 receptors as treatment targets in schizophrenia. Clin Schizophr Relat Psychoses. 2010 Apr;4(1):56-73. PMID 20643630
- [Background] Sundstrom Poromaa I, Comasco E, Georgakis MK, Skalkidou A. Sex differences in depression during pregnancy and the postpartum period. J Neurosci Res. 2017 Jan 2;95(1-2):719-730. doi: 10.1002/jnr.23859. PMID 27870443
- [Background] Wehrl HF, Sauter AW, Divine MR, Pichler BJ. Combined PET/MR: a technology becomes mature. J Nucl Med. 2015 Feb;56(2):165-8. doi: 10.2967/jnumed.114.150318. Epub 2015 Jan 15. PMID 25593114
- [Background] Bailey DL, Pichler BJ, Guckel B, Barthel H, Beer AJ, Bremerich J, Czernin J, Drzezga A, Franzius C, Goh V, Hartenbach M, Iida H, Kjaer A, la Fougere C, Ladefoged CN, Law I, Nikolaou K, Quick HH, Sabri O, Schafer J, Schafers M, Wehrl HF, Beyer T. Combined PET/MRI: Multi-modality Multi-parametric Imaging Is Here: Summary Report of the 4th International Workshop on PET/MR Imaging; February 23-27, 2015, Tubingen, Germany. Mol Imaging Biol. 2015 Oct;17(5):595-608. doi: 10.1007/s11307-015-0886-9. PMID 26286794
- [Background] Riedl V, Bienkowska K, Strobel C, Tahmasian M, Grimmer T, Forster S, Friston KJ, Sorg C, Drzezga A. Local activity determines functional connectivity in the resting human brain: a simultaneous FDG-PET/fMRI study. J Neurosci. 2014 Apr 30;34(18):6260-6. doi: 10.1523/JNEUROSCI.0492-14.2014. PMID 24790196
- [Background] Bailey DL, Antoch G, Bartenstein P, Barthel H, Beer AJ, Bisdas S, Bluemke DA, Boellaard R, Claussen CD, Franzius C, Hacker M, Hricak H, la Fougere C, Guckel B, Nekolla SG, Pichler BJ, Purz S, Quick HH, Sabri O, Sattler B, Schafer J, Schmidt H, van den Hoff J, Voss S, Weber W, Wehrl HF, Beyer T. Combined PET/MR: The Real Work Has Just Started. Summary Report of the Third International Workshop on PET/MR Imaging; February 17-21, 2014, Tubingen, Germany. Mol Imaging Biol. 2015 Jun;17(3):297-312. doi: 10.1007/s11307-014-0818-0. PMID 25672749
- [Background] Gilbert P, Allan S, Brough S, Melley S, Miles JN. Relationship of anhedonia and anxiety to social rank, defeat and entrapment. J Affect Disord. 2002 Sep;71(1-3):141-51. doi: 10.1016/s0165-0327(01)00392-5. PMID 12167510
- [Background] Etkin A, Egner T, Kalisch R. Emotional processing in anterior cingulate and medial prefrontal cortex. Trends Cogn Sci. 2011 Feb;15(2):85-93. doi: 10.1016/j.tics.2010.11.004. Epub 2010 Dec 16. PMID 21167765
- [Background] Watson D, Weber K, Assenheimer JS, Clark LA, Strauss ME, McCormick RA. Testing a tripartite model: I. Evaluating the convergent and discriminant validity of anxiety and depression symptom scales. J Abnorm Psychol. 1995 Feb;104(1):3-14. doi: 10.1037//0021-843x.104.1.3. PMID 7897050
- [Background] Calabrese WR, Rudick MM, Simms LJ, Clark LA. Development and validation of Big Four personality scales for the Schedule for Nonadaptive and Adaptive Personality--Second Edition (SNAP-2). Psychol Assess. 2012 Sep;24(3):751-63. doi: 10.1037/a0026915. Epub 2012 Jan 16. PMID 22250598
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kulkarni J, Riedel A, de Castella AR, Fitzgerald PB, Rolfe TJ, Taffe J, Burger H. Estrogen - a potential treatment for schizophrenia. Schizophr Res. 2001 Mar 1;48(1):137-44. doi: 10.1016/s0920-9964(00)00088-8. PMID 11278160
- [Background] Barch DM, Marder SR, Harms MP, Jarskog LF, Buchanan RW, Cronenwett W, Chen LS, Weiss M, Maguire RP, Pezous N, Feuerbach D, Lopez-Lopez C, Johns DR, Behrje RB, Gomez-Mancilla B. Task-related fMRI responses to a nicotinic acetylcholine receptor partial agonist in schizophrenia: A randomized trial. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Nov 3;71:66-75. doi: 10.1016/j.pnpbp.2016.06.013. Epub 2016 Jun 28. PMID 27371157
- [Background] Insel C, Reinen J, Weber J, Wager TD, Jarskog LF, Shohamy D, Smith EE. Antipsychotic dose modulates behavioral and neural responses to feedback during reinforcement learning in schizophrenia. Cogn Affect Behav Neurosci. 2014 Mar;14(1):189-201. doi: 10.3758/s13415-014-0261-3. PMID 24557585
- [Background] Jarskog LF, Dong Z, Kangarlu A, Colibazzi T, Girgis RR, Kegeles LS, Barch DM, Buchanan RW, Csernansky JG, Goff DC, Harms MP, Javitt DC, Keefe RS, McEvoy JP, McMahon RP, Marder SR, Peterson BS, Lieberman JA. Effects of davunetide on N-acetylaspartate and choline in dorsolateral prefrontal cortex in patients with schizophrenia. Neuropsychopharmacology. 2013 Jun;38(7):1245-52. doi: 10.1038/npp.2013.23. Epub 2013 Jan 16. PMID 23325325
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW + 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. Fertil Steril. 2012 Apr;97(4):843-51. doi: 10.1016/j.fertnstert.2012.01.128. Epub 2012 Feb 16. PMID 22341880
- [Background] Soules MR, Sherman S, Parrott E, Rebar R, Santoro N, Utian W, Woods N. Stages of Reproductive Aging Workshop (STRAW). J Womens Health Gend Based Med. 2001 Nov;10(9):843-8. doi: 10.1089/152460901753285732. PMID 11747678
- [Background] Franken IH, Rassin E, Muris P. The assessment of anhedonia in clinical and non-clinical populations: further validation of the Snaith-Hamilton Pleasure Scale (SHAPS). J Affect Disord. 2007 Apr;99(1-3):83-9. doi: 10.1016/j.jad.2006.08.020. Epub 2006 Sep 20. PMID 16996138
- [Background] Krystal AD, Pizzagalli DA, Smoski M, Mathew SJ, Nurnberger J Jr, Lisanby SH, Iosifescu D, Murrough JW, Yang H, Weiner RD, Calabrese JR, Sanacora G, Hermes G, Keefe RSE, Song A, Goodman W, Szabo ST, Whitton AE, Gao K, Potter WZ. A randomized proof-of-mechanism trial applying the 'fast-fail' approach to evaluating kappa-opioid antagonism as a treatment for anhedonia. Nat Med. 2020 May;26(5):760-768. doi: 10.1038/s41591-020-0806-7. Epub 2020 Mar 30. PMID 32231295
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Hafkenscheid A. Reliability of a standardized and expanded Brief Psychiatric Rating Scale: a replication study. Acta Psychiatr Scand. 1993 Nov;88(5):305-10. doi: 10.1111/j.1600-0447.1993.tb03464.x. PMID 8296573
- [Background] Keller J, Gomez RG, Kenna HA, Poesner J, DeBattista C, Flores B, Schatzberg AF. Detecting psychotic major depression using psychiatric rating scales. J Psychiatr Res. 2006 Feb;40(1):22-9. doi: 10.1016/j.jpsychires.2005.07.003. Epub 2005 Sep 13. PMID 16165160
- [Background] Coyle D, McGinnity TM, Prasad G. Creating a nonparametric brain-computer interface with neural time-series prediction preprocessing. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:2183-6. doi: 10.1109/IEMBS.2006.260626. PMID 17946502
- [Background] Pelizza L, Garlassi S, Azzali S, Paterlini F, Scazza I, Chiri LR, Poletti M, Pupo S, Raballo A. Anhedonia in young people with first episode psychosis: a longitudinal study. Nord J Psychiatry. 2020 Aug;74(6):381-389. doi: 10.1080/08039488.2020.1733661. Epub 2020 Feb 28. PMID 32108539
- [Background] Trostheim M, Eikemo M, Meir R, Hansen I, Paul E, Kroll SL, Garland EL, Leknes S. Assessment of Anhedonia in Adults With and Without Mental Illness: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Aug 3;3(8):e2013233. doi: 10.1001/jamanetworkopen.2020.13233. PMID 32789515
- [Background] Keller MB, Klein DN, Hirschfeld RM, Kocsis JH, McCullough JP, Miller I, First MB, Holzer CP 3rd, Keitner GI, Marin DB, et al. Results of the DSM-IV mood disorders field trial. Am J Psychiatry. 1995 Jun;152(6):843-9. doi: 10.1176/ajp.152.6.843. PMID 7755112
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Eckstrand KL, Forbes EE, Bertocci MA, Chase HW, Greenberg T, Lockovich J, Stiffler R, Aslam HA, Graur S, Bebko G, Phillips ML. Anhedonia Reduction and the Association Between Left Ventral Striatal Reward Response and 6-Month Improvement in Life Satisfaction Among Young Adults. JAMA Psychiatry. 2019 Sep 1;76(9):958-965. doi: 10.1001/jamapsychiatry.2019.0864. PMID 31066876
- [Background] Marder SR, Meibach RC. Risperidone in the treatment of schizophrenia. Am J Psychiatry. 1994 Jun;151(6):825-35. doi: 10.1176/ajp.151.6.825. PMID 7514366
- [Background] Yung AR, Phillips LJ, Yuen HP, Francey SM, McFarlane CA, Hallgren M, McGorry PD. Psychosis prediction: 12-month follow up of a high-risk ("prodromal") group. Schizophr Res. 2003 Mar 1;60(1):21-32. doi: 10.1016/s0920-9964(02)00167-6. PMID 12505135
- [Background] Watson D, O'Hara MW, Simms LJ, Kotov R, Chmielewski M, McDade-Montez EA, Gamez W, Stuart S. Development and validation of the Inventory of Depression and Anxiety Symptoms (IDAS). Psychol Assess. 2007 Sep;19(3):253-68. doi: 10.1037/1040-3590.19.3.253. PMID 17845118
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 2008 Sep-Oct;61(1-2):78-84. doi: 10.1016/j.maturitas.2008.09.011. PMID 19434881
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Gordon JL, Rubinow DR, Eisenlohr-Moul TA, Xia K, Schmidt PJ, Girdler SS. Efficacy of Transdermal Estradiol and Micronized Progesterone in the Prevention of Depressive Symptoms in the Menopause Transition: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):149-157. doi: 10.1001/jamapsychiatry.2017.3998. PMID 29322164
- [Background] Sarason IG, Johnson JH, Siegel JM. Assessing the impact of life changes: development of the Life Experiences Survey. J Consult Clin Psychol. 1978 Oct;46(5):932-46. doi: 10.1037//0022-006x.46.5.932. No abstract available. PMID 701572
- [Background] Lindenstruth KA, Curtis CB, Allen JK. Recruitment of African American and white postmenopausal women into clinical trials: the beneficial effects of soy trial experience. Ethn Dis. 2006 Autumn;16(4):938-42. PMID 17061750
- [Background] Knutson B, Fong GW, Bennett SM, Adams CM, Hommer D. A region of mesial prefrontal cortex tracks monetarily rewarding outcomes: characterization with rapid event-related fMRI. Neuroimage. 2003 Feb;18(2):263-72. doi: 10.1016/s1053-8119(02)00057-5. PMID 12595181
- [Background] Schultz W. Predictive reward signal of dopamine neurons. J Neurophysiol. 1998 Jul;80(1):1-27. doi: 10.1152/jn.1998.80.1.1. PMID 9658025
- [Background] Fischl B, Salat DH, Busa E, Albert M, Dieterich M, Haselgrove C, van der Kouwe A, Killiany R, Kennedy D, Klaveness S, Montillo A, Makris N, Rosen B, Dale AM. Whole brain segmentation: automated labeling of neuroanatomical structures in the human brain. Neuron. 2002 Jan 31;33(3):341-55. doi: 10.1016/s0896-6273(02)00569-x. PMID 11832223
- [Background] Knutson B, Fong GW, Adams CM, Varner JL, Hommer D. Dissociation of reward anticipation and outcome with event-related fMRI. Neuroreport. 2001 Dec 4;12(17):3683-7. doi: 10.1097/00001756-200112040-00016. PMID 11726774
- [Background] Crowther A, Smoski MJ, Minkel J, Moore T, Gibbs D, Petty C, Bizzell J, Schiller CE, Sideris J, Carl H, Dichter GS. Resting-state connectivity predictors of response to psychotherapy in major depressive disorder. Neuropsychopharmacology. 2015 Jun;40(7):1659-73. doi: 10.1038/npp.2015.12. Epub 2015 Jan 12. PMID 25578796
- [Background] Greene RK, Spanos M, Alderman C, Walsh E, Bizzell J, Mosner MG, Kinard JL, Stuber GD, Chandrasekhar T, Politte LC, Sikich L, Dichter GS. The effects of intranasal oxytocin on reward circuitry responses in children with autism spectrum disorder. J Neurodev Disord. 2018 Mar 27;10(1):12. doi: 10.1186/s11689-018-9228-y. PMID 29587625
- [Background] Choi EY, Yeo BT, Buckner RL. The organization of the human striatum estimated by intrinsic functional connectivity. J Neurophysiol. 2012 Oct;108(8):2242-63. doi: 10.1152/jn.00270.2012. Epub 2012 Jul 25. PMID 22832566
- [Background] Wang D, Liu H. Functional connectivity architecture of the human brain: not all the same. Neuroscientist. 2014 Oct;20(5):432-8. doi: 10.1177/1073858414543290. Epub 2014 Jul 16. PMID 25030990
- [Background] Whitfield-Gabrieli S, Nieto-Castanon A. Conn: a functional connectivity toolbox for correlated and anticorrelated brain networks. Brain Connect. 2012;2(3):125-41. doi: 10.1089/brain.2012.0073. Epub 2012 Jul 19. PMID 22642651
- [Background] Behzadi Y, Restom K, Liau J, Liu TT. A component based noise correction method (CompCor) for BOLD and perfusion based fMRI. Neuroimage. 2007 Aug 1;37(1):90-101. doi: 10.1016/j.neuroimage.2007.04.042. Epub 2007 May 3. PMID 17560126
- [Background] Koepp MJ, Gunn RN, Lawrence AD, Cunningham VJ, Dagher A, Jones T, Brooks DJ, Bench CJ, Grasby PM. Evidence for striatal dopamine release during a video game. Nature. 1998 May 21;393(6682):266-8. doi: 10.1038/30498. PMID 9607763
- [Background] Schott BH, Minuzzi L, Krebs RM, Elmenhorst D, Lang M, Winz OH, Seidenbecher CI, Coenen HH, Heinze HJ, Zilles K, Duzel E, Bauer A. Mesolimbic functional magnetic resonance imaging activations during reward anticipation correlate with reward-related ventral striatal dopamine release. J Neurosci. 2008 Dec 24;28(52):14311-9. doi: 10.1523/JNEUROSCI.2058-08.2008. PMID 19109512
- [Background] Sander CY, Hooker JM, Catana C, Rosen BR, Mandeville JB. Imaging Agonist-Induced D2/D3 Receptor Desensitization and Internalization In Vivo with PET/fMRI. Neuropsychopharmacology. 2016 Apr;41(5):1427-36. doi: 10.1038/npp.2015.296. Epub 2015 Sep 21. PMID 26388148
- [Background] Urban NB, Slifstein M, Meda S, Xu X, Ayoub R, Medina O, Pearlson GD, Krystal JH, Abi-Dargham A. Imaging human reward processing with positron emission tomography and functional magnetic resonance imaging. Psychopharmacology (Berl). 2012 May;221(1):67-77. doi: 10.1007/s00213-011-2543-6. Epub 2011 Nov 4. PMID 22052081
- [Background] Weiland BJ, Heitzeg MM, Zald D, Cummiford C, Love T, Zucker RA, Zubieta JK. Relationship between impulsivity, prefrontal anticipatory activation, and striatal dopamine release during rewarded task performance. Psychiatry Res. 2014 Sep 30;223(3):244-52. doi: 10.1016/j.pscychresns.2014.05.015. Epub 2014 Jun 5. PMID 24969539
- [Background] Lammertsma AA, Hume SP. Simplified reference tissue model for PET receptor studies. Neuroimage. 1996 Dec;4(3 Pt 1):153-8. doi: 10.1006/nimg.1996.0066. PMID 9345505
- [Background] Baker JH, Eisenlohr-Moul T, Wu YK, Schiller CE, Bulik CM, Girdler SS. Ovarian hormones influence eating disorder symptom variability during the menopause transition: A pilot study. Eat Behav. 2019 Dec;35:101337. doi: 10.1016/j.eatbeh.2019.101337. Epub 2019 Oct 25. PMID 31726420
- [Background] Eisenlohr-Moul TA, Rubinow DR, Schiller CE, Johnson JL, Leserman J, Girdler SS. Histories of abuse predict stronger within-person covariation of ovarian steroids and mood symptoms in women with menstrually related mood disorder. Psychoneuroendocrinology. 2016 May;67:142-52. doi: 10.1016/j.psyneuen.2016.01.026. Epub 2016 Feb 1. PMID 26896670
- [Background] Kinard JL, Mosner MG, Greene RK, Addicott M, Bizzell J, Petty C, Cernasov P, Walsh E, Eisenlohr-Moul T, Carter RM, McLamb M, Hopper A, Sukhu R, Dichter GS. Neural Mechanisms of Social and Nonsocial Reward Prediction Errors in Adolescents with Autism Spectrum Disorder. Autism Res. 2020 May;13(5):715-728. doi: 10.1002/aur.2273. Epub 2020 Feb 11. PMID 32043748
- [Background] Mosner MG, McLaurin RE, Kinard JL, Hakimi S, Parelman J, Shah JS, Bizzell J, Greene RK, Cernasov PM, Walsh E, Addicott MA, Eisenlohr-Moul T, Carter RM, Dichter GS. Neural Mechanisms of Reward Prediction Error in Autism Spectrum Disorder. Autism Res Treat. 2019 Jul 1;2019:5469191. doi: 10.1155/2019/5469191. eCollection 2019. PMID 31354993
- [Background] Walsh EC, Eisenlohr-Moul TA, Pedersen CA, Rubinow DR, Girdler SS, Dichter GS. Early Life Abuse Moderates the Effects of Intranasal Oxytocin on Symptoms of Premenstrual Dysphoric Disorder: Preliminary Evidence From a Placebo-Controlled Trial. Front Psychiatry. 2018 Nov 29;9:547. doi: 10.3389/fpsyt.2018.00547. eCollection 2018. PMID 30555357
- [Background] Kwapil TR. Social anhedonia as a predictor of the development of schizophrenia-spectrum disorders. J Abnorm Psychol. 1998 Nov;107(4):558-65. doi: 10.1037//0021-843x.107.4.558. PMID 9830243
- [Background] Wardenaar KJ, Giltay EJ, van Veen T, Zitman FG, Penninx BW. Symptom dimensions as predictors of the two-year course of depressive and anxiety disorders. J Affect Disord. 2012 Feb;136(3):1198-203. doi: 10.1016/j.jad.2011.11.037. Epub 2011 Dec 15. PMID 22177741
- [Background] Spijker J, Bijl RV, de Graaf R, Nolen WA. Determinants of poor 1-year outcome of DSM-III-R major depression in the general population: results of the Netherlands Mental Health Survey and Incidence Study (NEMESIS). Acta Psychiatr Scand. 2001 Feb;103(2):122-30. doi: 10.1034/j.1600-0447.2001.103002122.x. PMID 11167315
- [Background] McMakin DL, Olino TM, Porta G, Dietz LJ, Emslie G, Clarke G, Wagner KD, Asarnow JR, Ryan ND, Birmaher B, Shamseddeen W, Mayes T, Kennard B, Spirito A, Keller M, Lynch FL, Dickerson JF, Brent DA. Anhedonia predicts poorer recovery among youth with selective serotonin reuptake inhibitor treatment-resistant depression. J Am Acad Child Adolesc Psychiatry. 2012 Apr;51(4):404-11. doi: 10.1016/j.jaac.2012.01.011. Epub 2012 Mar 3. PMID 22449646
- [Background] Downar J, Geraci J, Salomons TV, Dunlop K, Wheeler S, McAndrews MP, Bakker N, Blumberger DM, Daskalakis ZJ, Kennedy SH, Flint AJ, Giacobbe P. Anhedonia and reward-circuit connectivity distinguish nonresponders from responders to dorsomedial prefrontal repetitive transcranial magnetic stimulation in major depression. Biol Psychiatry. 2014 Aug 1;76(3):176-85. doi: 10.1016/j.biopsych.2013.10.026. Epub 2013 Nov 28. PMID 24388670
- [Background] Keller J, Young CB, Kelley E, Prater K, Levitin DJ, Menon V. Trait anhedonia is associated with reduced reactivity and connectivity of mesolimbic and paralimbic reward pathways. J Psychiatr Res. 2013 Oct;47(10):1319-28. doi: 10.1016/j.jpsychires.2013.05.015. Epub 2013 Jun 19. PMID 23791396
- [Background] Treadway MT, Zald DH. Parsing Anhedonia: Translational Models of Reward-Processing Deficits in Psychopathology. Curr Dir Psychol Sci. 2013 Jun 1;22(3):244-249. doi: 10.1177/0963721412474460. PMID 24748727
- [Background] Pizzagalli DA, Iosifescu D, Hallett LA, Ratner KG, Fava M. Reduced hedonic capacity in major depressive disorder: evidence from a probabilistic reward task. J Psychiatr Res. 2008 Nov;43(1):76-87. doi: 10.1016/j.jpsychires.2008.03.001. Epub 2008 Apr 22. PMID 18433774
- [Background] Berridge KC, Kringelbach ML. Affective neuroscience of pleasure: reward in humans and animals. Psychopharmacology (Berl). 2008 Aug;199(3):457-80. doi: 10.1007/s00213-008-1099-6. Epub 2008 Mar 3. PMID 18311558
- [Background] Carl H, Walsh E, Eisenlohr-Moul T, Minkel J, Crowther A, Moore T, Gibbs D, Petty C, Bizzell J, Dichter GS, Smoski MJ. Sustained anterior cingulate cortex activation during reward processing predicts response to psychotherapy in major depressive disorder. J Affect Disord. 2016 Oct;203:204-212. doi: 10.1016/j.jad.2016.06.005. Epub 2016 Jun 4. PMID 27295377
- [Background] Schmidt PJ, Ben Dor R, Martinez PE, Guerrieri GM, Harsh VL, Thompson K, Koziol DE, Nieman LK, Rubinow DR. Effects of Estradiol Withdrawal on Mood in Women With Past Perimenopausal Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jul;72(7):714-26. doi: 10.1001/jamapsychiatry.2015.0111. PMID 26018333
- [Background] Santoro N, Epperson CN, Mathews SB. Menopausal Symptoms and Their Management. Endocrinol Metab Clin North Am. 2015 Sep;44(3):497-515. doi: 10.1016/j.ecl.2015.05.001. PMID 26316239
- [Background] Stewart DE, Boydell K, Derzko C, Marshall V. Psychologic distress during the menopausal years in women attending a menopause clinic. Int J Psychiatry Med. 1992;22(3):213-20. doi: 10.2190/EWRH-4P7E-ACMH-3MEN. PMID 1487384
- [Background] Robinson GE. Psychotic and mood disorders associated with the perimenopausal period: epidemiology, aetiology and management. CNS Drugs. 2001;15(3):175-84. doi: 10.2165/00023210-200115030-00002. PMID 11463126
- [Background] Schmidt PJ, Haq N, Rubinow DR. A longitudinal evaluation of the relationship between reproductive status and mood in perimenopausal women. Am J Psychiatry. 2004 Dec;161(12):2238-44. doi: 10.1176/appi.ajp.161.12.2238. PMID 15569895
- [Background] Yoest KE, Cummings JA, Becker JB. Estradiol, dopamine and motivation. Cent Nerv Syst Agents Med Chem. 2014;14(2):83-9. doi: 10.2174/1871524914666141226103135. PMID 25540977
- [Background] Yoest KE, Quigley JA, Becker JB. Rapid effects of ovarian hormones in dorsal striatum and nucleus accumbens. Horm Behav. 2018 Aug;104:119-129. doi: 10.1016/j.yhbeh.2018.04.002. Epub 2018 Apr 22. PMID 29626485
- [Background] Chavez C, Hollaus M, Scarr E, Pavey G, Gogos A, van den Buuse M. The effect of estrogen on dopamine and serotonin receptor and transporter levels in the brain: an autoradiography study. Brain Res. 2010 Mar 19;1321:51-9. doi: 10.1016/j.brainres.2009.12.093. Epub 2010 Jan 14. PMID 20079719
- [Background] Brzezinski A, Brzezinski-Sinai NA, Seeman MV. Treating schizophrenia during menopause. Menopause. 2017 May;24(5):582-588. doi: 10.1097/GME.0000000000000772. PMID 27824682
- [Background] Dichter GS, Felder JN, Petty C, Bizzell J, Ernst M, Smoski MJ. The effects of psychotherapy on neural responses to rewards in major depression. Biol Psychiatry. 2009 Nov 1;66(9):886-97. doi: 10.1016/j.biopsych.2009.06.021. Epub 2009 Sep 2. PMID 19726030
- [Background] Walsh EC, Eisenlohr-Moul TA, Minkel J, Bizzell J, Petty C, Crowther A, Carl H, Smoski MJ, Dichter GS. Pretreatment brain connectivity during positive emotion upregulation predicts decreased anhedonia following behavioral activation therapy for depression. J Affect Disord. 2019 Jan 15;243:188-192. doi: 10.1016/j.jad.2018.09.065. Epub 2018 Sep 17. PMID 30245249
- [Background] Walsh E, Carl H, Eisenlohr-Moul T, Minkel J, Crowther A, Moore T, Gibbs D, Petty C, Bizzell J, Smoski MJ, Dichter GS. Attenuation of Frontostriatal Connectivity During Reward Processing Predicts Response to Psychotherapy in Major Depressive Disorder. Neuropsychopharmacology. 2017 Mar;42(4):831-843. doi: 10.1038/npp.2016.179. Epub 2016 Sep 2. PMID 27585739
- [Background] Willi J, Ehlert U. Assessment of perimenopausal depression: A review. J Affect Disord. 2019 Apr 15;249:216-222. doi: 10.1016/j.jad.2019.02.029. Epub 2019 Feb 11. PMID 30776662
- [Background] Rubinow DR, Schmidt PJ. Is there a role for reproductive steroids in the etiology and treatment of affective disorders? Dialogues Clin Neurosci. 2018 Sep;20(3):187-196. doi: 10.31887/DCNS.2018.20.3/drubinow. PMID 30581288
- [Background] Seeman MV, Gonzalez-Rodriguez A. Use of psychotropic medication in women with psychotic disorders at menopause and beyond. Curr Opin Psychiatry. 2018 May;31(3):183-192. doi: 10.1097/YCO.0000000000000410. PMID 29528895
- [Background] Schiller CE, Minkel J, Smoski MJ, Dichter GS. Remitted major depression is characterized by reduced prefrontal cortex reactivity to reward loss. J Affect Disord. 2013 Nov;151(2):756-762. doi: 10.1016/j.jad.2013.06.016. Epub 2013 Jul 5. PMID 23835103
- [Derived] Walsh MJM, Gibson K, Hynd M, Eisenlohr-Moul TA, Walsh EC, Schiff L, Jarskog F, Lalush D, Dichter GS, Schiller CE. Perimenopausal Effects of Estradiol on Anhedonia and Psychosis Study (PEEPs): study protocol for a neural and molecular mechanistic clinical trial. Trials. 2023 Feb 28;24(1):150. doi: 10.1186/s13063-023-07166-7. PMID 36855177